CLINICAL TRIAL: NCT05720728
Title: Research of New Serological Markers for the Diagnosis and Monitoring of Candidaemia in Hospitalized Patients
Acronym: 2419
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 2419
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Candida Infection
MeSH Terms: conditions — Candidiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: collection of blood samples — For each patient, a serum sample collected at the time when candidemia is suspected (time of execution of blood cultures) will be examined. For patients with candidemia, all serum samples taken during infection follow-up will also be examined.

SUMMARY:
Bloodstream infections due to Candida spp remain a serious medical challenge because of their high incidence and poor outcome. Diagnosis and monitoring of patients are still problematic, hindering efficient clinical management of the disease. The invastigators propose here to perform a retrospective study in a clinically well-characterized candidemic patient, with the goal of recognizing host immunological factors and virulence-associated fungal molecules relevant in the onset and evolution of infection. The researchers' ultimate goal is to identify new diagnostic and/or prognostic benchmarks useful in clinical settings. By combining serologic and immunologic expertise with clinical expertise, the research team has real potential to generate new markers of host pathogenesis and immune response in candidemia and to inform prospective clinical trials to control this terrible disease

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized
* one or more positive blood cultures for Candida spp,
* positive beta-glucanemia
* the presence of at least one clinical symptom of infection will be considered cases of candidemia.

Exclusion Criteria:

* age less than 18 years
* state of immunosuppression
* incompleteness of clinical data
* unavailability of serum samples in sufficient quantities for analysis and in good condition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients hospitalized one or more positive blood cultures for Candida spp, positive beta-glucanemia and the presence of at least one clinical symptom of infection will be considered cases of candidemia.
  Controls will be defined as patients at risk of candidaemia but with negative blood cultures and who have never started antifungal therapy in the 30 days following the date of the 1st blood culture.
  Patients at risk are defined as patients with fever who have at least two of the following factors: CVC, parenteral nutrition, antibiotic therapy in the previous 30 days for at least 7 days, abdominal surgery, polytrauma, dialysis, diabetes, at least two sites colonized by Candida.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
levels of antibodies | 1 year
  i) presence and levels of antibodies directed towards beta-glucans and Candida virulence proteins.
  ii) presence and levels of circulating Candida virulence proteins. iii) presence and levels of soluble mediators of innate immunity and inflammation No genetic analysis will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione PoliclinicoAgostino Gemelli IRCCS, Rome, Roma, Italy